CLINICAL TRIAL: NCT03398941
Title: The Effect of Preoperative Long Period Octreotide Combined With Postoperative Short Period Octreotide on the Complications After Pancreatectomy. A Prospective, Multicenter Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengfeng Wang (Other)
Responsible Party: Sponsor-Investigator, Chengfeng Wang, Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC2017L01
Record Dates: First submitted 2018-01-07; First posted 2018-01-16 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: Pancreatic Diseases
Keywords: Pancreatic fistula
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined group (Experimental)
  Interventions: Drug: Preoperative Long Period Octreotide Combined With Postoperative Short Period Octreotide

INTERVENTIONS:
Drug: Preoperative Long Period Octreotide Combined With Postoperative Short Period Octreotide — Long-Period Octreotide 20mg one week before operation combine Short Period Octreotide 0.3mg during postoperative five days.

SUMMARY:
The Effect of Preoperative Long Period Octreotide Combined With Postoperative Short Period Octreotide on the Complications After Pancreatectomy. A Prospective, Multicenter Clinical Trial

DETAILED DESCRIPTION:
The trial is funded by Cancer Foundation of China. The trial is prepared to be registered on the clinicaltrail.gov.

Quality assurance plan: every participant is enrolled or excluded by two practiced investigators. And two investigators participated in all steps of the trail, including the record of the data, and the investigators will compare the data. If the data is consistent, the investigators would record the data; if not, the data would be checked and decided by the two investigators. All the steps and data are site monitored and audited by the workers of research and financial department of National Cancer Center/ Cancer Hospital, Chinese Academy of Medical Sciences.

Data check: the investigators compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry. Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources, including medical records and electronic case report forms.

Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information, and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as participants recruitment, data collection, data management, data analysis, reporting for adverse events, and change management. All registry operations would be done according to specific steps, and by two practiced investigators.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect. According to the formula to differ advantages and disadvantages, the investigators need at least 70 participants to take part in the trail.

The investigators can recruit about 150 participants according to previous experiences.

Plan for missing data: the investigators would collect as much data as possible, and the investigators exclude the participants who cannot cooperate on recruitment. And the investigators manage situations according to statistical principles where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results.

Statistical analysis plan: Kaplan-Meier method would be used to analyze the difference of survival time between the two groups, and the local control rate of the two groups would be compared by chi square test. Statistical analyses would be performed by using IBM SPSS Statistics(version 20; IBM, Chicago, USA). The level of significance is defined as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatectomy patients

Exclusion Criteria:

* Treated by chemotherapy or radiotherapy before With distant organ metastasis Cannot tolerate surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
pancreatic fistula | three week after operation
delayed gastric emptying | three week after operation
intra-abdominal fluid collections | three week after operation
wound infection | three week after operation
Bile leak | three week after operation
Abdominal bleeding | three week after operation

CONTACTS AND LOCATIONS:
Overall Officials: Wang Chengfeng, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No